CLINICAL TRIAL: NCT05578261
Title: Explore the Impacts of One Session Theta Burst Stimulation Over Cerebellum in Adults With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202200409A0
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (Experimental): All of the participants will accept one session iTBS over right Crus I/II. The total pulses of every session are 1200 pulses (600 pulses with 15 minutes interval)
  *iTBS = intermittent theta burst stimulation.
  Interventions: Device: intermittent theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — stimulatory protocol

SUMMARY:
The investigator would like to investigate the impact of theta-burst stimulation over cerebellum in adults with autism spectrum disorder

ELIGIBILITY:
Inclusion Criteria:

* Adults with autism spectrum disorder (≥18 years old), confirmed by Autism Diagnostic Observation Schedule.

Exclusion Criteria:

* Previous or current severe neurological disorder such as epilepsy, visual or hearing impairment.
* Previous or current severe systemic disease such as cardiovascular disease, diabetes or infection.
* Previous or current severe brain injury
* Implementation of metal materials such as pacemaker or medication pump
* Previous or current severe psychiatric disorders such as schizophrenia, bipolar disorder or substance abuse
* Pregnancy
* Individuals with a significant brain abnormality such as intracranial space occupied lesions
* History of brain surgery or nervous system infection, such as meningitis and encephalitis
* Concurrent use of medications which increased the risk of seizure attack
* Participate another clinical trial within one month
* Skin trauma on application site
* Individuals suffering from multiple sclerosis
* Individuals with a large ischemic scar
* Individuals suffering from sleep deprivation during rTMS procedures
* Individuals with a heavy consumption of alcohol
* Current taking antiepileptic drugs
* Individuals with a migraine headache from increased intracranial pressure
* Unable to complete MRI scan

Withdrawal criteria:

* Seizure attack during study period
* Autistic symptoms worsened obviously during study period
* Extreme agitation or irritability during study period
* Participants request
* Take antiepileptic drug during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Adverse effects report form (Headache) | 1 week after iTBS (post iTBS)
  Recording adverse effects in participants after iTBS.
Adverse effects report form (Dizziness) | 1 week after iTBS (post iTBS)
  Recording adverse effects in participants after iTBS.
Adverse effects report form (Tinnitus) | 1 week after iTBS (post iTBS)
  Recording adverse effects in participants after iTBS.
Adverse effects report form (Seizure) | 1 week after iTBS (post iTBS)
  Recording adverse effects in participants after iTBS.
Adverse effects report form (Other) | 1 week after iTBS (post iTBS)
  Recording adverse effects in participants after iTBS.

SECONDARY OUTCOMES:
MRI T1 | Within one month
  Brain structural volumes (cm²)
functional MRI (resting-state/biological motion task) - BOLD signal | Within one month
  Blood-oxygen-level-dependent (BOLD) signal is a measurement used in fMRI, which reflects the neural activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan